CLINICAL TRIAL: NCT03897595
Title: A Multi-centre, Prospective Post Marketing Surveillance Study to Assess Mid-term Performance of the Mpact Cup in Subjects Requiring Primary Total Hip Arthroplasty
Brief Title: Assess the Mid-term Performance of the Mpact Cup in Subjects Requiring Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.014.08/01
Record Dates: First submitted 2019-03-11; First posted 2019-04-01 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Mpact cup: Quadra®-H, Quadra®-C, AMIStem®-H or AMIStem®-C femoral stem and Mpact® Acetabular hip system with CoCr Femoral Head or Ceramic MectaCer BIOLOX® Femoral Head
  Interventions: Device: MPact Cup

INTERVENTIONS:
Device: MPact Cup — Quadra®-H, Quadra®-C, AMIStem®-H or AMIStem®-C femoral stem and Mpact® Acetabular hip system with CoCr Femoral Head or Ceramic MectaCer BIOLOX® Femoral Head

SUMMARY:
Monitor the performance of the Mpact cup in the treatment of patients with hip joint disease requiring a total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to the patient's surgery.

  * Those presenting with disease that meets the indications for use for Medacta USA implants defined by this study (on-label use).
  * Patients must be willing to comply with the pre and post-operative evaluation schedule

Exclusion Criteria:

* Those with one or more medical conditions identified as a contraindication defined by the labeling on any Medacta implants used in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Harris Hip Scores (HHS) | Pre-operative, 3 or 6 months, 1 year, 2 year and 5 year
  Assessment of improvement of clinical outcomes following total hip replacement surgery using the Harris Hip Scores
Change from baseline of implant survivorship | Post-operative 3 or 6 months, 1 year, 2 year, and 5 year
  Assessment of bone fracture, implant fracture, neck reabsorption
Change in baseline of Complications | Day of surgery, post-operative 3 or 6 months, 1 year, 2 year, and 5 year.
  Assessment of Adverse events and serious adverse events
Change in baseline fixation and wear | Post-operative 3 or 6 months, 1 year, 2 year and 5 year
  Radiographic analysis by measuring Radio Lucent Lines
Change in baseline fixation | Post-operative 3 or 6 months, 1 year, 2 year and 5 year
  Radiographic analysis by measuring implant fixation in millimeters

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Denver Vail Orthopedics, Parker, Colorado
  - Saint Alphonsus Medical Group, Boise, Idaho
  - Illinois Bone and Joint Institute, Libertyville, Illinois
  - McBride Orthopedic Hospital, Oklahoma City, Oklahoma
  - Jordan Valley Medical Center of Orthopedics Rehabilitation and Excellence, West Jordan, Utah